CLINICAL TRIAL: NCT02624869
Title: Open-label, Single-Arm, Multicenter Study to Evaluate the Safety, Tolerability and Efficacy of Evolocumab for LDL-C Reduction, as Add-on to Diet and Lipid-lowering Therapy, in Pediatric Subjects From 10 to 17 Years of Age With Heterozygous Familial Hypercholesterolemia (HeFH) or Homozygous Familial Hypercholesterolemia (HoFH)
Brief Title: Safety, Tolerability and Efficacy of Evolocumab (AMG 145) in Children With Inherited Elevated Low-density Lipoprotein Cholesterol (Familial Hypercholesterolemia)
Acronym: HAUSER-OLE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20120124; 2015-002276-25 (EudraCT Number)
Record Dates: First submitted 2015-10-22; First posted 2015-12-09 (Estimated); Results first posted 2022-01-14 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Familial Hypercholesterolemia
Keywords: Hypercholesterolemia; Elevated Cholesterol; High Cholesterol; PCSK9 mutations; Severe Familial Hypercholesterolemia; evolocumab; Repatha; Heterozygous Familial Hypercholesterolemia; Homozygous Familial Hypercholesterolemia; Pediatric; Paediatric
MeSH Terms: conditions — Hyperlipoproteinemia Type II; Hypercholesterolemia; Homozygous Familial Hypercholesterolemia | interventions — evolocumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Evolocumab (Experimental): Participants receive 420 mg evolocumab administered by subcutaneous injection every 4 weeks (QM) for up to 80 weeks.
  Interventions: Biological: Evolocumab

INTERVENTIONS:
Biological: Evolocumab — Administered by subcutaneous injection
  Other Names: Repatha®; AMG 145

SUMMARY:
The main purpose of this study is to describe the safety and tolerability of 80 weeks of subcutaneous (SC) evolocumab when added to standard of care in children 10 to 17 years of age with familial hypercholesterolemia.

ELIGIBILITY:
Inclusion Criteria:

Heterozygous Familial Hypercholesterolemia (HeFH):

-Completed Study 20120123 (NCT02392559) while still on assigned investigational product and did not experience a treatment-related serious adverse event

Homozygous Familial Hypercholesterolemia (HoFH):

* Male or female, ≥ 10 to ≤ 17 years of age at time of enrollment
* Diagnosis of HoFH
* On a low-fat diet and receiving background lipid-lowering therapy
* Lipid-lowering therapy unchanged for ≥ 4 weeks prior to LDL-C screening; fibrates must be stable for at least 6 weeks prior to screening.
* Fasting LDL-C at screening ≥ 130 mg/dL (3.4 mmol/L)
* Fasting triglycerides ≤ 400 mg/dL (4.5 mmol/L)

Exclusion Criteria:

-Currently receiving treatment in another investigational device or drug study, or less than 30 days since ending treatment on another investigational device or drug study(s); except Study 20120123

HoFH:

* Moderate to severe renal dysfunction
* Active liver disease or hepatic dysfunction,
* Creatine kinase > 3 times the upper limit of normal (ULN) at screening

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 163 (Actual)
Dates: Start 2016-09-10 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (43):
- United States (3):
  - Research Site, The Bronx, New York
  - Research Site, Cincinnati, Ohio
  - Research Site, Nashville, Tennessee
- Research Site, Camperdown, New South Wales, Australia
- Austria (3):
  - Research Site, Feldkirch
  - Research Site, Salzburg
  - Research Site, Vienna
- Belgium (3):
  - Research Site, Ghent
  - Research Site, La Louvière
  - Research Site, Leuven
- Brazil (3):
  - Research Site, Fortaleza, Ceará
  - Research Site, Brasília, Federal District
  - Research Site, São Paulo
- Canada (2):
  - Research Site, Chicoutimi, Quebec
  - Research Site, Québec, Quebec
- Colombia (2):
  - Research Site, Barranquilla, Atlántico
  - Research Site, Bucaramanga, Santander Department
- Research Site, Svitavy, Czechia
- Greece (2):
  - Research Site, Athens
  - Research Site, Thessaloniki
- Research Site, Budapest, Hungary
- Italy (4):
  - Research Site, Palermo
  - Research Site, Pisa
  - Research Site, Roma
  - Research Site, Torino
- Research Site, Kota Bharu, Kelantan, Malaysia
- Research Site, Amsterdam, Netherlands
- Norway (2):
  - Research Site, Bergen
  - Research Site, Oslo
- Research Site, Gdansk, Poland
- Research Site, Guimarães, Portugal
- Research Site, Saint Petersburg, Russia
- Research Site, Ljubljana, Slovenia
- South Africa (2):
  - Research Site, Parktown, Gauteng
  - Research Site, Parow, Western Cape
- Spain (3):
  - Research Site, Córdoba, Andalusia
  - Research Site, A Coruña, Galicia
  - Research Site, Lugo, Galicia
- Switzerland (2):
  - Research Site, Geneva
  - Research Site, Reinach
- Turkey (Türkiye) (2):
  - Research Site, Ankara
  - Research Site, Izmir
- Research Site, Birmingham, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the link below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- [Background] Santos RD, Ruzza A, Hovingh GK, Stefanutti C, Mach F, Descamps OS, Bergeron J, Wang B, Bartuli A, Buonuomo PS, Greber-Platzer S, Luirink I, Bhatia AK, Raal FJ, Kastelein JJP, Wiegman A, Gaudet D. Paediatric patients with heterozygous familial hypercholesterolaemia treated with evolocumab for 80 weeks (HAUSER-OLE): a single-arm, multicentre, open-label extension of HAUSER-RCT. Lancet Diabetes Endocrinol. 2022 Oct;10(10):732-740. doi: 10.1016/S2213-8587(22)00221-2. Epub 2022 Sep 5. PMID 36075246
- [Background] Raal FJ, Hegele RA, Ruzza A, Lopez JAG, Bhatia AK, Wu J, Wang H, Gaudet D, Wiegman A, Wang J, Santos RD. Evolocumab Treatment in Pediatric Patients With Homozygous Familial Hypercholesterolemia: Pooled Data From Three Open-Label Studies. Arterioscler Thromb Vasc Biol. 2024 May;44(5):1156-1164. doi: 10.1161/ATVBAHA.123.320268. Epub 2024 Mar 28. PMID 38545781
- [Background] Santos RD, Ruzza A, Wang B, Maruff P, Schembri A, Bhatia AK, Mach F, Bergeron J, Gaudet I, St Pierre J, Kastelein JJP, Hovingh GK, Wiegman A, Gaudet D, Raal FJ. Evolocumab in paediatric heterozygous familial hypercholesterolaemia: cognitive function during 80 weeks of open-label extension treatment. Eur J Prev Cardiol. 2024 Feb 15;31(3):302-310. doi: 10.1093/eurjpc/zwad332. PMID 37855448
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 46 centers in 23 countries (Australia, Austria, Belgium, Brazil, Canada, Colombia, Czech Republic, Greece, Hungary, Italy, Malaysia, Netherlands, Norway, Poland, Portugal, Russia, Slovenia, South Africa, Spain, Switzerland, Turkey, United Kingdom, and United States of America).
Pre-assignment Details: This study enrolled participants with heterozygous familial hypercholesterolemia (HeFH) who had completed the parent study 20120123 (NCT02392559) without experiencing a treatment-related serious adverse event, and children 10 to 17 years of age with a diagnosis of homozygous familial hypercholesterolemia (HoFH).
Groups:
- HeFH (Placebo in Parent Study): Evolocumab 420 mg QM: Participants with heterozygous familial hypercholesterolemia (HeFH) who had received placebo in the parent study received 420 mg evolocumab administered by subcutaneous injection every 4 weeks (QM) for up to 80 weeks.
- HeFH (Evolocumab in Parent Study): Evolocumab 420 mg QM: Participants with HeFH who had received evolocumab in the parent study received 420 mg evolocumab administered by subcutaneous injection every 4 weeks for up to 80 weeks.
- HoFH: Evolocumab 420 mg QM: Participants with homozygous familial hypercholesterolemia (HoFH) received 420 mg evolocumab administered by subcutaneous injection every 4 weeks for up to 80 weeks.
Period: Overall Study
Arm/Group | HeFH (Placebo in Parent Study): Evolocumab 420 mg QM | HeFH (Evolocumab in Parent Study): Evolocumab 420 mg QM | HoFH: Evolocumab 420 mg QM
Started | 49 | 101 | 13
Received Study Drug | 49 | 101 | 12
Completed | 48 | 98 | 11
Not Completed | 1 | 3 | 2
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 3 | 1

BASELINE CHARACTERISTICS:
Population: All enrolled participants
Groups:
- HeFH (Placebo in Parent Study): Evolocumab 420 mg QM: Participants with HeFH who had received placebo in the parent study received 420 mg evolocumab administered by subcutaneous injection every 4 weeks (QM) for up to 80 weeks.
- HoFH: Evolocumab 420 mg QM: Participants with HoFH received 420 mg evolocumab administered by subcutaneous injection every 4 weeks for up to 80 weeks.
- Total: Total of all reporting groups
Arm/Group | HeFH (Placebo in Parent Study): Evolocumab 420 mg QM | HeFH (Evolocumab in Parent Study): Evolocumab 420 mg QM | HoFH: Evolocumab 420 mg QM | Total
Number analyzed (Participants) | 49 | 101 | 13 | 163
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.8 (2.5) | 14.2 (2.4) | 12.4 (2.0) | 14.0 (2.5)
Age, Customized [Count of Participants; unit: Participants] — Eight HeFH participants were 18 years old at the time of rollover into Study 20120124, however all were ≤ 17 years old at the time of enrollment into the parent study 20120123.
  Participants
    2 - 11 years | 11 | 18 | 6 | 35
    12 - 17 years | 37 | 76 | 7 | 120
    18 - 64 years | 1 | 7 | 0 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 59 | 2 | 85
  Male | 25 | 42 | 11 | 78
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 6 | 0 | 13
  Not Hispanic or Latino | 42 | 95 | 13 | 150
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 2 | 2 | 4
  Black or African American | 0 | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  White | 40 | 86 | 9 | 135
  Other | 9 | 11 | 2 | 22
Region [Count of Participants; unit: Participants]
  North America | 8 | 12 | 0 | 20
  Europe | 33 | 65 | 7 | 105
  Latin America | 8 | 18 | 0 | 26
  Asia Pacific | 0 | 6 | 6 | 12
Low-density Lipoprotein Cholesterol (LDL-C) Concentration [Mean (Standard Deviation); unit: mg/dL] — For participants with HeFH who rolled over from parent study 20120123, baseline values are defined as parent study baseline concentrations; for de novo participants with HoFH, baseline values are defined as the mean of the two most recent non-missing concentrations measured through the central laboratory prior to or on Study Day 1. Population: The full analysis set included all participants with HeFH from parent Study 20120123 who were enrolled and dosed as well as all participants with HoFH who were enrolled and dosed in this study.
  mg/dL
    number analyzed (Participants) | 49 | 101 | 12 | 162
    (all) | 184.0 (48.3) | 184.4 (45.2) | 426.0 (166.4) | 202.2 (88.8)
Non-High-Density Lipoprotein Cholesterol (Non-HDL-C) Concentration [Mean (Standard Deviation); unit: mg/dL] — For participants with HeFH who rolled over from parent study 20120123, baseline values are defined as parent study baseline concentrations; for de novo participants with HoFH, baseline values are defined as the mean of the two most recent non-missing concentrations measured through the central laboratory prior to or on Study Day 1. Population: Full analysis set
  mg/dL
    number analyzed (Participants) | 49 | 101 | 12 | 162
    (all) | 201.0 (49.3) | 203.4 (47.5) | 443.7 (170.8) | 220.5 (90.2)
Apolipoprotein B (ApoB) Concentration [Mean (Standard Deviation); unit: mg/dL] — For participants with HeFH who rolled over from parent study 20120123, baseline values are defined as parent study baseline concentrations; for de novo participants with HoFH, baseline values are defined as the mean of the two most recent non-missing concentrations measured through the central laboratory prior to or on Study Day 1. Population: Full analysis set with available baseline data
  mg/dL
    number analyzed (Participants) | 47 | 100 | 12 | 159
    (all) | 119.1 (28.1) | 123.1 (27.4) | 250.1 (84.9) | 131.5 (48.6)
Total Cholesterol/High-density Lipoprotein Cholesterol (HDL-C) Ratio [Mean (Standard Deviation); unit: ratio] — For participants with HeFH who rolled over from parent study 20120123, baseline values are defined as parent study baseline concentrations; for de novo participants with HoFH, baseline values are defined as the mean of the two most recent non-missing concentrations measured through the central laboratory prior to or on Study Day 1. Population: Full analysis set with available baseline data
  ratio
    number analyzed (Participants) | 49 | 101 | 12 | 162
    (all) | 5.546 (1.541) | 5.716 (1.809) | 14.707 (7.891) | 6.331 (3.557)
Apolipoprotein B/Apolipoprotein A1 Ratio [Mean (Standard Deviation); unit: ratio] — For participants with HeFH who rolled over from parent study 20120123, baseline values are defined as parent study baseline concentrations; for de novo participants with HoFH, baseline values are defined as the mean of the two most recent non-missing concentrations measured through the central laboratory prior to or on Study Day 1. Population: Full analysis set with available baseline data
  ratio
    number analyzed (Participants) | 47 | 100 | 12 | 159
    (all) | 0.943 (0.265) | 0.972 (0.306) | 2.388 (1.036) | 1.070 (0.545)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event is defined as any untoward medical occurrence in a clinical trial participant, not necessarily having a causal relationship with study treatment.
  A serious AE is as an AE that met at least 1 of the following criteria:
  * fatal;
  * life threatening;
  * required in-patient hospitalization or prolongation of existing hospitalization;
  * resulted in persistent or significant disability/incapacity;
  * congenital anomaly/birth defect;
  * other medically important serious event.
  AEs were graded for severity using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0:
  Grade 1: Mild; asymptomatic or mild symptoms; Grade 2: Moderate; minimal, local or noninvasive intervention indicated; Grade 3: Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; Grade 4: Life-threatening consequences; urgent intervention indicated; Grade 5: Death related to AE.
Time Frame: From first dose of evolocumab in this study up to and including 30 days after the last dose or up to the end of study date, whichever was earlier; up to 80 weeks.
Population: Full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | HeFH (Placebo in Parent Study): Evolocumab 420 mg QM | HeFH (Evolocumab in Parent Study): Evolocumab 420 mg QM | HoFH: Evolocumab 420 mg QM
Number analyzed (Participants) | 49 | 101 | 12
Participants
  Any treatment-emergent adverse event (TEAE) | 36 | 69 | 7
  TEAE ≥ Grade 2 | 25 | 56 | 5
  TEAE ≥ Grade 3 | 4 | 2 | 2
  TEAE ≥ Grade 4 | 0 | 1 | 0
  Serious adverse events | 2 | 2 | 2
  TEAE leading to discontinuation of evolocumab | 0 | 0 | 0
  Fatal adverse events | 0 | 0 | 0

2. Secondary Outcome: Percent Change From Baseline to Week 80 in Low-density Lipoprotein Cholesterol (LDL-C) in HeFH Participants
Description: For HeFH participants baseline was defined as the baseline value of the parent study 20120123.
Time Frame: Baseline and week 80
Population: Full analysis set with available data
Measure: Mean (Standard Error); unit: percent change
Arm/Group | HeFH (Placebo in Parent Study): Evolocumab 420 mg QM | HeFH (Evolocumab in Parent Study): Evolocumab 420 mg QM
Number analyzed (Participants) | 40 | 88
percent change | -36.01 (4.28) | -34.96 (3.05)

3. Secondary Outcome: Percent Change From Baseline to Week 80 in Low-density Lipoprotein Cholesterol (LDL-C) in HoFH Participants
Description: For HoFH participants baseline was defined as the baseline value in this study (20120124).
Time Frame: Baseline and week 80
Population: Full analysis set with available data
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | HoFH: Evolocumab 420 mg QM
Number analyzed (Participants) | 11
percent change | -14.29 [-40.61 to 3.54]

4. Secondary Outcome: Percent Change From Baseline to Week 80 in Non-HDL-C in HeFH Participants
Description: For HeFH participants baseline was defined as the baseline value of the parent study 20120123.
Time Frame: Baseline and week 80
Population: Full analysis set with available data
Measure: Mean (Standard Error); unit: percent change
Arm/Group | HeFH (Placebo in Parent Study): Evolocumab 420 mg QM | HeFH (Evolocumab in Parent Study): Evolocumab 420 mg QM
Number analyzed (Participants) | 40 | 88
percent change | -32.37 (3.96) | -31.95 (2.89)

5. Secondary Outcome: Percent Change From Baseline to Week 80 in Non-HDL-C in HoFH Participants
Description: For HoFH participants baseline was defined as the baseline value in this study (20120124).
Time Frame: Baseline and week 80
Population: Full analysis set with available data
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | HoFH: Evolocumab 420 mg QM
Number analyzed (Participants) | 11
percent change | -13.03 [-40.68 to 2.69]

6. Secondary Outcome: Percent Change From Baseline to Week 80 in Apolipoprotein B in HeFH Participants
Description: For HeFH participants baseline was defined as the baseline value in the parent study 20120123.
Time Frame: Baseline and week 80
Population: Full analysis set with available data
Measure: Mean (Standard Error); unit: percent change
Arm/Group | HeFH (Placebo in Parent Study): Evolocumab 420 mg QM | HeFH (Evolocumab in Parent Study): Evolocumab 420 mg QM
Number analyzed (Participants) | 44 | 87
percent change | -27.10 (3.32) | -24.15 (2.99)

7. Secondary Outcome: Percent Change From Baseline to Week 80 in Apolipoprotein B in HoFH Participants
Description: For HoFH participants baseline was defined as the baseline value in this study (20120124).
Time Frame: Baseline and week 80
Population: Full analysis set with available data
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | HoFH: Evolocumab 420 mg QM
Number analyzed (Participants) | 11
percent change | -19.17 [-33.33 to 11.59]

8. Secondary Outcome: Percent Change From Baseline to Week 80 in Total Cholesterol/HDL-C Ratio in HeFH Participants
Description: For HeFH participants baseline was defined as the baseline value in the parent study 20120123.
Time Frame: Baseline and week 80
Population: Full analysis set with available data
Measure: Mean (Standard Error); unit: percent change
Arm/Group | HeFH (Placebo in Parent Study): Evolocumab 420 mg QM | HeFH (Evolocumab in Parent Study): Evolocumab 420 mg QM
Number analyzed (Participants) | 40 | 88
percent change | -28.78 (3.48) | -28.32 (2.47)

9. Secondary Outcome: Percent Change From Baseline to Week 80 in Total Cholesterol/HDL-C Ratio in HoFH Participants
Description: For HoFH participants baseline was defined as the baseline value in this study (20120124).
Time Frame: Baseline and week 80
Population: Full analysis set with available data
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | HoFH: Evolocumab 420 mg QM
Number analyzed (Participants) | 11
percent change | 3.71 [-41.17 to 7.57]

10. Secondary Outcome: Percent Change From Baseline to Week 80 in Apolipoprotein B / Apolipoprotein A1 Ratio in HeFH Participants
Description: For HeFH participants baseline was defined as the baseline value in the parent study 20120123.
Time Frame: Baseline and week 80
Population: Full analysis set with available data
Measure: Mean (Standard Error); unit: percent change
Arm/Group | HeFH (Placebo in Parent Study): Evolocumab 420 mg QM | HeFH (Evolocumab in Parent Study): Evolocumab 420 mg QM
Number analyzed (Participants) | 44 | 87
percent change | -31.00 (3.66) | -29.89 (2.80)

11. Secondary Outcome: Percent Change From Baseline to Week 80 in Apolipoprotein B/Apolipoprotein A1 Ratio in HoFH Participants
Description: For HoFH participants baseline was defined as the baseline value in this study (20120124).
Time Frame: Baseline and week 80
Population: Full analysis set with available data
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | HoFH: Evolocumab 420 mg QM
Number analyzed (Participants) | 11
percent change | -2.96 [-35.71 to 9.30]

12. Secondary Outcome: Change From Baseline to Week 80 in LDL-C in HeFH Participants
Description: For HeFH participants baseline was defined as the baseline value of the parent study 20120123.
Time Frame: Baseline and week 80
Population: Full analysis set with available data
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | HeFH (Placebo in Parent Study): Evolocumab 420 mg QM | HeFH (Evolocumab in Parent Study): Evolocumab 420 mg QM
Number analyzed (Participants) | 40 | 88
mg/dL | -67.2 (8.2) | -63.1 (5.6)

13. Secondary Outcome: Change From Baseline to Week 80 in LDL-C in HoFH Participants
Description: For HoFH participants baseline was defined as the baseline value in this study (20120124).
Time Frame: Baseline and week 80
Population: Full analysis set with available data
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | HoFH: Evolocumab 420 mg QM
Number analyzed (Participants) | 11
mg/dL | -36.5 [-180.5 to 16.0]

14. Secondary Outcome: Change From Baseline to Week 80 in Estradiol Levels
Description: For HeFH participants baseline was defined as the baseline value in the parent study 20120123. For HoFH participants baseline was defined as the baseline value in this study (20120124).
Time Frame: Baseline and week 80
Population: Full analysis set; female participants with available data
Measure: Mean (Standard Error); unit: pmol/L
Arm/Group | HeFH (Placebo in Parent Study): Evolocumab 420 mg QM | HeFH (Evolocumab in Parent Study): Evolocumab 420 mg QM | HoFH: Evolocumab 420 mg QM
Number analyzed (Participants) | 23 | 54 | 2
pmol/L | 131.3 (45.3) | 48.2 (58.1) | 283.0 (130.0)

15. Secondary Outcome: Change From Baseline to Week 80 in Testosterone Levels
Description: as for outcome 14
Time Frame: Baseline and week 80
Population: Full analysis set; male participants with available data
Measure: Mean (Standard Error); unit: nmol/L
Arm/Group | HeFH (Placebo in Parent Study): Evolocumab 420 mg QM | HeFH (Evolocumab in Parent Study): Evolocumab 420 mg QM | HoFH: Evolocumab 420 mg QM
Number analyzed (Participants) | 18 | 34 | 7
nmol/L | 5.282 (1.567) | 3.230 (1.167) | 2.916 (0.984)

16. Secondary Outcome: Change From Baseline to Week 80 in Follicle Stimulating Hormone (FSH) Levels
Description: as for outcome 14
Time Frame: Baseline and week 80
Population: Full analysis set with available data
Measure: Mean (Standard Error); unit: IU/L
Arm/Group | HeFH (Placebo in Parent Study): Evolocumab 420 mg QM | HeFH (Evolocumab in Parent Study): Evolocumab 420 mg QM | HoFH: Evolocumab 420 mg QM
Number analyzed (Participants) | 44 | 91 | 10
IU/L | 1.88 (0.90) | 0.60 (0.37) | 1.18 (0.35)

17. Secondary Outcome: Change From Baseline to Week 80 in Luteinizing Hormone (LH) Levels
Description: as for outcome 14
Time Frame: Baseline and week 80
Population: Full analysis set with available data
Measure: Mean (Standard Error); unit: IU/L
Arm/Group | HeFH (Placebo in Parent Study): Evolocumab 420 mg QM | HeFH (Evolocumab in Parent Study): Evolocumab 420 mg QM | HoFH: Evolocumab 420 mg QM
Number analyzed (Participants) | 44 | 92 | 10
IU/L | 2.88 (1.51) | 1.04 (0.95) | 1.76 (0.84)

18. Secondary Outcome: Change From Baseline to Week 80 in Adenocorticotropic Hormone (ACTH) Levels
Description: as for outcome 14
Time Frame: Baseline and week 80
Population: Full analysis set with available data
Measure: Mean (Standard Error); unit: pmol/L
Arm/Group | HeFH (Placebo in Parent Study): Evolocumab 420 mg QM | HeFH (Evolocumab in Parent Study): Evolocumab 420 mg QM | HoFH: Evolocumab 420 mg QM
Number analyzed (Participants) | 43 | 84 | 11
pmol/L | 0.78 (0.55) | 0.55 (0.61) | -0.75 (1.79)

19. Secondary Outcome: Change From Baseline to Week 80 in Dehydroepiandrosterone Sulfate (DHEA-S) Levels
Description: as for outcome 14
Time Frame: Baseline and week 80
Population: Full analysis set with available data
Measure: Mean (Standard Error); unit: μmol/L
Arm/Group | HeFH (Placebo in Parent Study): Evolocumab 420 mg QM | HeFH (Evolocumab in Parent Study): Evolocumab 420 mg QM | HoFH: Evolocumab 420 mg QM
Number analyzed (Participants) | 43 | 89 | 11
μmol/L | 1.051 (0.222) | 0.956 (0.126) | 0.944 (0.247)

20. Secondary Outcome: Change From Baseline to Week 80 in Cortisol Levels
Description: as for outcome 14
Time Frame: Baseline and week 80
Population: Full analysis set with available data
Measure: Mean (Standard Error); unit: nmol/L
Arm/Group | HeFH (Placebo in Parent Study): Evolocumab 420 mg QM | HeFH (Evolocumab in Parent Study): Evolocumab 420 mg QM | HoFH: Evolocumab 420 mg QM
Number analyzed (Participants) | 43 | 90 | 11
nmol/L | 29.81 (28.34) | 51.18 (25.19) | 57.26 (56.11)

21. Secondary Outcome: Number of Participants With Liver Function Test Abnormalities at Week 80
Description: Liver function tests included alanine aminotransferase (ALT) levels, aspartate aminotransferase (AST) levels and total bilirubin levels.
Time Frame: Week 80
Population: Full analysis set with available data at week 80
Measure: Count of Participants; unit: Participants
Arm/Group | HeFH (Placebo in Parent Study): Evolocumab 420 mg QM | HeFH (Evolocumab in Parent Study): Evolocumab 420 mg QM | HoFH: Evolocumab 420 mg QM
Number analyzed (Participants) | 45 | 91 | 10
Participants
  ALT or AST > 3 x ULN | 0 | 0 | 0
  ALT or AST > 5 x ULN | 0 | 0 | 0
  Total bilirubin > 2 x ULN | 0 | 2 | 1

22. Secondary Outcome: Number of Participants With Abnormalities in Levels of Creatine Kinase (CK) at Week 80
Description: The number of participants with levels of creatine kinase greater than 5 times the upper limit of normal (ULN) and greater than 10 times the ULN, measured by the central laboratory.
Time Frame: Week 80
Population: Full analysis set with available data at week 80
Measure: Count of Participants; unit: Participants
Arm/Group | HeFH (Placebo in Parent Study): Evolocumab 420 mg QM | HeFH (Evolocumab in Parent Study): Evolocumab 420 mg QM | HoFH: Evolocumab 420 mg QM
Number analyzed (Participants) | 45 | 90 | 10
Participants
  CK > 5 x ULN | 0 | 0 | 1
  CK > 10 x ULN | 0 | 0 | 0

23. Secondary Outcome: Change From Baseline to Week 80 in Carotid Intima-media Thickness (cIMT)
Description: Carotid intima-media thickness measures the thickness of the intima and media, the inner two layers of the carotid artery, and is used to determine the extent of plaque buildup in the walls of the arteries (atherosclerosis) supplying blood to the head.
  CIMT was measured by ultrasonography and analyzed at a core laboratory. The largest values measured in the left common carotid artery (LCCA) and the right common carotid artery (RCCA) are averaged in this analysis.
Time Frame: Baseline and week 80
Population: Full analysis set with available data
Measure: Mean (Standard Error); unit: mm
Arm/Group | HeFH (Placebo in Parent Study): Evolocumab 420 mg QM | HeFH (Evolocumab in Parent Study): Evolocumab 420 mg QM | HoFH: Evolocumab 420 mg QM
Number analyzed (Participants) | 34 | 59 | 7
mm | -0.019 (0.007) | -0.012 (0.006) | 0.006 (0.032)

24. Secondary Outcome: Change From Baseline in Height at Weeks 24, 48, and 80
Time Frame: Baseline and weeks 24, 48, and 80
Population: Full analysis set with available data at each time point.
Measure: Mean (Standard Error); unit: cm
Arm/Group | HeFH (Placebo in Parent Study): Evolocumab 420 mg QM | HeFH (Evolocumab in Parent Study): Evolocumab 420 mg QM | HoFH: Evolocumab 420 mg QM
Number analyzed (Participants) | 49 | 101 | 12
cm
  Females: Baseline: number analyzed (Participants) | 24 | 59 | 2
  Females: Baseline | 158.1 (2.3) | 157.9 (1.3) | 149.4 (7.1)
  Females: Change at week 24: number analyzed (Participants) | 21 | 55 | 2
  Females: Change at week 24 | 2.8 (0.7) | 2.0 (0.4) | 1.6 (1.1)
  Females: Change at week 48: number analyzed (Participants) | 22 | 55 | 2
  Females: Change at week 48 | 4.2 (1.0) | 2.8 (0.5) | 1.4 (2.4)
  Females: Change at week 80: number analyzed (Participants) | 24 | 56 | 2
  Females: Change at week 80 | 4.0 (1.7) | 3.4 (0.7) | 2.4 (3.9)
  Males: Baseline: number analyzed (Participants) | 25 | 42 | 10
  Males: Baseline | 158.2 (3.0) | 163.7 (1.9) | 158.9 (4.8)
  Males: Change at week 24: number analyzed (Participants) | 23 | 40 | 10
  Males: Change at week 24 | 3.4 (0.5) | 3.8 (0.5) | 3.8 (0.8)
  Males: Change at week 48: number analyzed (Participants) | 23 | 39 | 9
  Males: Change at week 48 | 6.2 (0.8) | 6.2 (0.7) | 5.3 (1.2)
  Males: Change at week 80: number analyzed (Participants) | 21 | 36 | 9
  Males: Change at week 80 | 9.3 (1.5) | 9.0 (1.1) | 9.2 (1.6)

25. Secondary Outcome: Change From Baseline in Weight at Weeks 24, 48, and 80
Time Frame: Baseline and weeks 24, 48, and 80
Population: Full analysis set with available data at each time point
Measure: Mean (Standard Error); unit: kg
Arm/Group | HeFH (Placebo in Parent Study): Evolocumab 420 mg QM | HeFH (Evolocumab in Parent Study): Evolocumab 420 mg QM | HoFH: Evolocumab 420 mg QM
Number analyzed (Participants) | 49 | 101 | 12
kg
  Females: Baseline: number analyzed (Participants) | 24 | 59 | 2
  Females: Baseline | 52.8 (2.9) | 57.0 (2.0) | 42.7 (1.3)
  Females: Change at week 24: number analyzed (Participants) | 21 | 55 | 2
  Females: Change at week 24 | 3.3 (0.8) | 2.3 (0.6) | 3.4 (2.1)
  Females: Change at week 48: number analyzed (Participants) | 22 | 54 | 2
  Females: Change at week 48 | 4.3 (1.1) | 3.5 (0.7) | 4.7 (5.3)
  Females: Change at week 80: number analyzed (Participants) | 24 | 56 | 2
  Females: Change at week 80 | 5.6 (1.3) | 5.2 (0.8) | 5.5 (4.2)
  Males: Baseline: number analyzed (Participants) | 25 | 42 | 10
  Males: Baseline | 54.1 (3.6) | 61.0 (3.2) | 51.7 (4.9)
  Males: Change at week 24: number analyzed (Participants) | 23 | 40 | 10
  Males: Change at week 24 | 4.4 (0.9) | 4.6 (0.7) | 4.6 (0.9)
  Males: Change at week 48: number analyzed (Participants) | 23 | 39 | 9
  Males: Change at week 48 | 6.8 (1.3) | 7.4 (1.0) | 7.6 (1.2)
  Males: Change at week 80: number analyzed (Participants) | 21 | 36 | 9
  Males: Change at week 80 | 10.9 (1.6) | 11.2 (1.4) | 10.6 (2.3)

26. Secondary Outcome: Number of Participants With Change in Tanner Staging From Baseline to Week 80
Description: Pubertal growth and sexual maturity was assessed separately for males and females using the 5 Tanner stages where stage 1 = prepubertal and stage 5 = mature.
  The number of participants with any change in Tanner Stage from baseline is reported.
Time Frame: Baseline and week 80
Population: Full analysis set with available data
Measure: Count of Participants; unit: Participants
Arm/Group | HeFH (Placebo in Parent Study): Evolocumab 420 mg QM | HeFH (Evolocumab in Parent Study): Evolocumab 420 mg QM | HoFH: Evolocumab 420 mg QM
Number analyzed (Participants) | 45 | 91 | 11
Participants
  Males: Staging by genital size: number analyzed (Participants) | 21 | 36 | 9
  Males: Staging by genital size | 13 | 20 | 6
  Males: Staging by pubic hair: number analyzed (Participants) | 21 | 36 | 9
  Males: Staging by pubic hair | 14 | 21 | 6
  Females: Staging by breast development: number analyzed (Participants) | 24 | 55 | 2
  Females: Staging by breast development | 11 | 27 | 1
  Females: Staging by pubic hair: number analyzed (Participants) | 24 | 55 | 2
  Females: Staging by pubic hair | 11 | 26 | 1

ADVERSE EVENTS:
Time Frame: From first dose of evolocumab in this study up to and including 30 days after the last dose or up to the end of study date, whichever was earlier; up to 80 weeks.
Description: Serious adverse events and other adverse events are reported for all participants who received at least one dose of study drug.
Arm/Group | HeFH (Placebo in Parent Study): Evolocumab 420 mg QM | HeFH (Evolocumab in Parent Study): Evolocumab 420 mg QM | HoFH: Evolocumab 420 mg QM
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/101 | 0/13
Serious Adverse Events (participants affected / at risk) | 2/49 | 2/101 | 2/12
Other Adverse Events (participants affected / at risk) | 27/49 | 45/101 | 7/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HeFH (Placebo in Parent Study): Evolocumab 420 mg QM (N=49) | HeFH (Evolocumab in Parent Study): Evolocumab 420 mg QM (N=101) | HoFH: Evolocumab 420 mg QM (N=12)
Appendicitis (Infections and infestations) | 0 | 0 | 1
Appendicitis perforated (Infections and infestations) | 1 | 0 | 0
Peritonitis (Infections and infestations) | 1 | 0 | 0
Arteriovenous fistula aneurysm (Injury, poisoning and procedural complications) | 0 | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0
Anorexia nervosa (Psychiatric disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | HeFH (Placebo in Parent Study): Evolocumab 420 mg QM (N=49) | HeFH (Evolocumab in Parent Study): Evolocumab 420 mg QM (N=101) | HoFH: Evolocumab 420 mg QM (N=12)
Abdominal pain upper (Gastrointestinal disorders) | 1 | 5 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 1
Fatigue (General disorders) | 4 | 3 | 0
Influenza like illness (General disorders) | 5 | 8 | 0
Injection site erythema (General disorders) | 4 | 1 | 0
Injection site haemorrhage (General disorders) | 0 | 1 | 1
Pyrexia (General disorders) | 5 | 1 | 0
Gastroenteritis (Infections and infestations) | 3 | 7 | 0
Influenza (Infections and infestations) | 0 | 3 | 1
Nasopharyngitis (Infections and infestations) | 8 | 14 | 0
Otitis media (Infections and infestations) | 0 | 1 | 1
Tonsillitis (Infections and infestations) | 0 | 4 | 1
Upper respiratory tract infection (Infections and infestations) | 3 | 6 | 1
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 | 0 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 3 | 1
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Headache (Nervous system disorders) | 4 | 9 | 1
Attention deficit hyperactivity disorder (Psychiatric disorders) | 2 | 2 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 5 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2020-05-27): https://cdn.clinicaltrials.gov/large-docs/69/NCT02624869/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-29): https://cdn.clinicaltrials.gov/large-docs/69/NCT02624869/SAP_001.pdf